CLINICAL TRIAL: NCT04834778
Title: A Multicenter, Open-label, Phase 1a Study of HC-5404-FU in Subjects With Advanced Solid Tumors
Brief Title: A Study of HC-5404-FU to Establish the Maximum Tolerated Dose (MTD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HC-404-FCP-2011
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Renal Cell Carcinoma; Gastric Cancer; Metastatic Breast Cancer; Small-cell Lung Cancer; Other Solid Tumors
Keywords: RCC; GC; MCA; SCLC; Phase 1; First in human; HC-5404-FU; HC-5404
MeSH Terms: conditions — Carcinoma, Renal Cell; Stomach Neoplasms; Breast Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 - 25 mg (Experimental): 25 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 2 - 50 mg (Experimental): 50 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 3 - 100 mg (Experimental): 100 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 4 - 200 mg (Experimental): 200 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 5 - 400 mg (Experimental): 400 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 6 - 600 mg (Experimental): 600 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 7 - 900 mg (Experimental): 900 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU
- Cohort 8 - 300 mg (Experimental): 300 mg capsules of HC-5404-FU administered orally twice a day with food or within 30 minutes of completing a meal of each 3-week treatment cycle
  Interventions: Drug: HC-5404-FU

INTERVENTIONS:
Drug: HC-5404-FU — HC 5404-FU (hemi fumarate salt of HC 5404) is a novel, highly selective, and potent PERK inhibitor. Preclinical pharmacological studies demonstrated high specificity of HC 5404-FU to PERK and decreased viability of tumor cells. HC 5404-FU will be orally administered BID every day with food or within 30 minutes of completing a meal, starting at 25 mg, with doses escalating to 50, 100, 200, 400, 600, and 900 mg BID as safety allows for each 3-week treatment cycle.
  Other Names: HC-5404

SUMMARY:
Study HC-404-FCP-2011 is a first in human, Phase 1a, multi-center, open-label study to establish the maximum tolerated dose (MTD) and evaluate the safety and tolerability of oral dosing of HC-5404-FU in a dose-escalating fashion. Up to 36 qualified subjects at 3 to 5 US sites, who have specific tumor types of renal cell carcinoma (RCC), gastric cancer (GC), metastatic breast cancer (MBC), small cell lung cancer (SCLC), and other solid tumors (e.g., non-small cell lung cancer, colorectal cancer, carcinoma of unknown primary) with the exception of rapidly progressing neoplasms (e.g., pancreatic cancer, glioblastoma, hepatocellular carcinoma) will receive HC-5404-FU. Every effort will be made to ensure approximately 50% of all subjects enrolled will be subjects with RCC and GC. The starting dose level is 25 mg twice daily (BID), escalating to 50, 100, and 200 mg BID as safety allows, following the Bayesian Optimal Interval (BOIN) design. The safety monitoring committee (SMC) will evaluate the DLTs and cumulative safety and PK data at the end of each cohort. Based on the SMC recommendations after a comprehensive review of PK and safety data for 200 mg BID dose, higher dose levels will be evaluated, starting with 400 mg BID. The dose will escalate to 600 mg and then 900 mg following the BOIN design starting with 1 subject at each escalated dose, until the MTD is reached or the sponsor or SMC declares the dose most appropriate for clinical development. This Phase 1a will be expanded into a Phase 1b/2a study through a protocol amendment and will then assess the dose and tumor type(s) selected in Phase 1a as the most appropriate for further clinical development. Subjects will be dosed until unacceptable toxicity, disease progression per immune-related Response Evaluation Criteria in Solid Tumors (iRECIST), subject withdrawal, any other administrative reasons, or after 2 years of treatment, whichever occurs first. Efficacy will be assessed via Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1); computed tomography (CT) scans will be conducted every 6 weeks. Safety, including occurrence of dose-limiting toxicities (DLTs), pharmacokinetics (PK), and biomarker parameters will also be assessed.

DETAILED DESCRIPTION:
HC 5404-FU will be orally administered BID with food or within 30 minutes of completing a meal, starting at 25 mg, with doses escalating to 50, 100, 200, 400, 600 and 900 mg BID as safety allows. Up to 24 subjects will be enrolled to ensure 12 subjects complete the study at the estimated MTD of HC 5404-FU. Dosing will occur in 3-week cycles. Subjects are to spend Cycle 1/Day 1 (C1D1) in the clinic followed by an overnight stay for safety monitoring and PK sampling. Subjects will be hospitalized for administration of first 3 doses: C1D1 am and pm doses, and Cycle 1/Day 2 (C1D2) am dose; on Days 8, 15, and 21 the am dose will be taken in the clinic after the planned PK samples. All other doses are to be self administered at home. After the initial hospital stay at the start of study, subjects will be seen in outpatient clinic on Days 8, 15, and 21 of Cycle 1 for PK assessment and thereafter, the first day of each cycle for physical and laboratory assessments, adverse event (AE), and dosing compliance monitoring; the end of treatment visit will also be in person in outpatient clinic.

Following completion of the treatment period of the study, subjects will be monitored for survival up for up to 24 months after the last post treatment follow-up visit.

Dose escalation will follow the Bayesian Optimal Interval (BOIN) design. The decision to escalate to the next dose level will be based on safety assessments after all subjects of a cohort have reached the end of Cycle 1/Day 21 (DLT evaluation period). The safety monitoring committee (SMC) will be responsible for dose escalation decisions, including whether to modify the dose escalation based on the DLT observations and review of available PK data.

The target toxicity rate of 30%, with limits of 0.236 to 0.359 for escalation/de escalation, will be employed to determine the MTD. With these predefined parameters, when the observed toxicity rate in a dose level is less than 0.236, the dose for the next cohort can escalate. If the observed toxicity rate is higher than 0.359, the dose will de escalate. Otherwise, the dose remains the same.

Individual subjects may be considered for treatment at a higher dose than the dose to which they were initially assigned after subject has completed 2 cycles of treatment and 1 postbaseline CT scan and maintained at least a stable disease (SD) response. In order to escalate a dose level, the subject must have tolerated his/her current dose level without experiencing a DLT, and the dose level to which the subject is planned to be escalated must have completed a DLT evaluation period, not exceeded the MTD, and been declared safe. Each subject can go through 2 dose escalations and do not need to go through a DLT evaluation period for either escalation. Intrasubject dose escalation will be considered on a case-by-case basis, each case to be assessed and approved by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Have a signed informed consent form prior to any study specific procedures or treatment
2. Be ≥18 years of age (male or female) at the time of consent
3. Have 1 of the following histologically or cytologically confirmed tumor types with qualifying characteristics, and have received a minimum of 2 (and no more than 5) lines of prior therapy for metastatic (Stage IV) disease:

   1. RCC (renal cell carcinoma - clear cell or papillary)
   2. SCLC (small cell lung cancer) OR have received a minimum of 3 (and no more than 5) lines of prior therapy for metastatic (Stage IV) disease:
   3. GC (gastric adenocarcinoma)
   4. Human epidermal growth factor receptor positive (HER2+) MBC (metastatic breast cancer)
   5. Other solid tumors (e.g., non-small cell lung cancer, colorectal cancer, carcinoma of unknown primary) with the exception of rapidly progressing neoplasms (e.g., pancreatic cancer, glioblastoma, hepatocellular carcinoma)

   Note: Subjects with RCC and GC are a priority and should constitute approximately 50% (12 subjects) of the enrolled popululation. Enrollment of all others will be capped when reaching a combined 50%, in order to maintain 12 slots for subjects with RCC and GC.
4. Have at least 1 radiologically measurable lesion as per RECIST v 1.1, defined as a lesion that is at least 10 mm in longest diameter or lymph node and that is at least 15 mm in short axis imaged by CT scan or magnetic resonance imaging (MRI) and obtained by imaging within 28 days prior to screening. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
5. Have resolution of all previous treatment related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (≤ Grade 2) and alopecia. If the subject received major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention
6. Provided there are suitable and accessible lesions, no biopsy contraindications, minimal risk of complications and a positive informed decision, subject as are willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality, for assessment of biomarker status. Two biopsies will be necessary: at baseline (within 30 days prior to first dose) and within 7 days after Cycle 3/Day 1.

   Newly obtained biopsy specimens are preferred to archived samples and formalin- fixed, paraffin-embedded block specimens are preferred to slides. In the event a fresh pre-treatment biopsy is not able to be provided, the most recent archival biopsy must be provided in its place
7. Have Eastern Cooperative Oncology Group performance status of 0 or 1 and sustained between screening and initiation of dosing on Day 1
8. QT interval corrected for heart rate using Fridericia's (QTcF) method ≤450 msec
9. Have an albumin level of ≥3 g/dL at screening
10. Have life expectancy of 3 months or greater as determined by the treating physician
11. Have adequate organ function within 15 days prior to first administration of study drug on Day 1, as defined by meeting all of the following criteria:

    1. Total bilirubin ≤1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5 x ULN
    2. Aspartate aminotransferase and alanine aminotransferase ≤2.5 × ULN or ≤5 × ULN for subjects with known hepatic metastases
    3. Fasting serum glucose within normal range and hemoglobin A1c ≤8%
    4. Thyroid function tests (thyroid stimulating hormone [TSH] within normal limits for subjects with normal thyroid function and free thyroxine [FT4]) within normal limits for subjects on thyroid treatment
12. Have adequate renal function within 15 days prior to first administration of study drug on Day 1, as defined by creatinine ≤1.5 × ULN and creatinine clearance ≥30 mL/min, as per the below Cockcroft Gault formula
13. Have adequate hematologic function within 15 days prior to first administration of study drug on Day 1, as defined by meeting all of the following criteria:

    1. Hemoglobin ≥9 g/dL (uncorrected by red blood cell transfusion or erythropoietin support)
    2. Absolute neutrophil count ≥1.5 × 109/L
    3. Platelet count ≥100 × 109/L
14. Have adequate coagulation function within 15 days prior to first administration of study drug on Day 1, as defined by either of the following criteria:

    1. International normalized ratio (INR) <1.5 × ULN OR for subjects receiving warfarin or low molecular weight heparin, the subject must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy
    2. Activated partial thromboplastin time (aPTT) <1.5 × ULN unless subject is receiving anticoagulant therapy, provided prothrombin time or aPTT is within therapeutic range of intended use of anticoagulants
15. Female subject of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
16. Female subject of childbearing potential must be willing to use an adequate form of contraception from the first dose of study medication through 90 days after the last dose of study drug
17. Female subject must agree not to breastfeed and not to donate ova starting at screening and throughout the study treatment, and for 90 days after the last dose of study drug
18. Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or for the time partner is breastfeeding throughout the study period and for 90 days after the last dose of study drug
19. Male subject with female partner(s) of childbearing potential must not donate sperm during the treatment period and for at least 90 days after the last dose of study drug
20. Male subject with female partner(s) of childbearing potential should agree to use a highly effective method of contraception during the treatment period and for at least 90 days after the last dose of the study drug
21. Be willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of study treatment or who has not recovered from adverse reactions due to a previously administered agent or major surgery
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
3. Has a diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids (≤30 mg/day of hydrocortisone, ≤10 mg/day of prednisone, ≤2 mg/day of dexamethasone, or equivalent) may be approved after consultation with the sponsor
4. Has taken a medication that is a strong CYP3A4 inhibitor or inducer within 4 weeks of the first dose of treatment (see Appendix 12)
5. Has known history of active tuberculosis
6. Has known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
7. Has known active Hepatitis B (anti hepatitis B surface antibody, anti hepatitis B core antibody, hepatitis B surface antigen [HBsAg]) or Hepatitis C (hepatitis C antibody) infection
8. Has a current diagnosis of severe acute respiratory syndrome coronavirus (SARS CoV) 2 infection confirmed by reverse transcription polymerase chain reaction (PCR) test. Subject needs to have a negative PCR test at screening and a negative PCR test within 14 days prior to the first dose of study treatment
9. Has a history of clinically severe autoimmune disease, or a history of organ transplant
10. Has insulin dependent (Type I) diabetes or poorly controlled Type II diabetes (per clinical discretion) with hemoglobin A1c >8%
11. Has known additional malignancy that is progressing or required active treatment within previous 5 years. Exceptions include basal cell carcinoma or squamous cell carcinoma of the skin that has undergone potentially curative therapy, superficial bladder cancer, or in situ cervical cancer. Subjects with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease free for at least 5 years
12. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of disease progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using systemic steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
13. Has a history of interstitial lung disease, pneumonitis within 12 months prior to screening or current pneumonitis
14. Has an active infection requiring systemic therapy
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
16. Has a history or ongoing clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome, symptomatic or uncontrolled arrhythmia, congestive heart failure, baseline ECG abnormalities, including, but not limited to, QTc prolongation (prolonged QTcF defined as ≥450 msec) or any Class III or IV cardiac disease as defined by the New York Heart Association Functional Classification
17. Has overt or latent disorders of the exocrine pancreas (such as acute or chronic pancreatitis of any etiology) or chronic (including autoimmune) gastrointestinal disorders such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, lupus, scleroderma, Sjogren's syndrome, and polyarteritis nodosa
18. Has a known psychiatric or substance abuse disorder(s) that would interfere with informed consent or cooperation with the requirements of the trial
19. Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the trial, starting with the prescreening or screening visit through 90 days after the last dose of study drug
20. Is a first degree relative of the investigator, staff, or study sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Determination of MTD of HC-5404-FU | Within 18 months of last patient enrolled
  When orally administered in a dose escalating fashion in subjects with selected, advanced solid tumors
Occurrence of dose-limiting toxicities (DLTs) | Within 18 months of last patient enrolled
Incidence and severity of treatment-emergent adverse events (TEAEs) and treatment related TEAEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 5.0 | Within 18 months of last patient enrolled
Incidence of TEAEs leading to premature discontinuation | Within 18 months of last patient enrolled
Incidence of significant laboratory abnormalities, based on hematology, serum chemistry, and urinalysis test results | Within 18 months of last patient enrolled
Incidence of abnormalities observed in 12 lead ECG parameters | Within 18 months of last patient enrolled
Incidence of abnormalities observed in vital signs measurements and physical examinations | Within 18 months of last patient enrolled

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 until last measurable concentration (AUC0 last) | Within 24 months of last patient enrolled
Area under the plasma concentration versus time curve from time 0 to 12 hours postdose (AUC0 12) | Within 24 months of last patient enrolled
Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0 ∞) | Within 24 months of last patient enrolled
Area under the plasma concentration versus time curve over a dosing interval (AUC0 t) | Within 24 months of last patient enrolled
Peak plasma concentration (Cmax) | Within 24 months of last patient enrolled
Time of the maximum observed plasma concentration (tmax) | Within 24 months of last patient enrolled
Apparent total clearance (CL/F) of plasma concentration | Within 24 months of last patient enrolled
Apparent volume of distribution during the terminal phase (Vz/F) of plasma concentration | Within 24 months of last patient enrolled
Apparent terminal elimination half life (t1/2) of plasma concentration | Within 24 months of last patient enrolled
Accumulation ratio based on AUC0 t (ARAUC) of plasma concentration | Within 24 months of last patient enrolled
Linearity ratio (LR) of plasma concentration | Within 24 months of last patient enrolled
Overall response rate (ORR) to HC-5404-FU using iRECIST | Within 24 months of last patient enrolled
Duration of response (DOR) to HC-5404-FU using iRECIST | Within 24 months of last patient enrolled
Time to treatment failure (TTF) | Within 24 months of last patient enrolled
Progression-free survival (PFS) using iRECIST | Within 24 months of last patient enrolled
Overall response (OS) using iRECIST | Within 24 months of last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Jose Iglesias, MD, Study Director — Consultant Chief Medical Officer for HiberCell, Inc.
Locations (4):
- United States (4):
  - Karmanos Cancer Institute, Detroit, Michigan
  - HealthPartners Cancer Care Center, Saint Paul, Minnesota
  - Baylor University Medical Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No